CLINICAL TRIAL: NCT07374692
Title: Observational Study of Responses to Treatments in Advanced Central Nervous System (CNS) Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10002539; 002539-C
Record Dates: First submitted 2026-01-28; First posted 2026-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Recurrent CNS Tumors; Brain Cancer; Gliomas; IDH-wildtype Gliomas; IDH-mutant Gliomas; Rare CNS Tumor
Keywords: CNS Tumor; Brain Tumor; Rare Tumor; SmartMatch; Gliomas; Drug Screen
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/SmartMatch testing (Other): Turnaround time for SmartMatch platform implementation and molecular profiling of recurrent CNS tumors
  Interventions: Other: Tumor sample collection

INTERVENTIONS:
Other: Tumor sample collection — Fresh tumor samples will be collected for the study only if available following a planned biopsy or resection performed at NIH.

SUMMARY:
Background:

Primary central nervous system (CNS) tumors grow in the brain and spinal cord. These tumors are rare, but they are difficult to treat and often fatal. SmartMatch is a new technology that tries to help find the best medicines for the particular tumor by testing how small pieces of surgically removed tumor tissue react to different drugs. The study team wants to see if SmartMatch can complete the analysis and generate a report within 21 days from the time of the surgery.

Objective:

To better understand CNS tumors so doctors can find better ways to treat them in the future.

Eligibility:

People aged 15 years and older with recurrent CNS tumors. Patient must already be scheduled for a surgery for the tumor at the NIH.

Design:

The study team will collect a small amount of tumor samples during the planned surgery. They may also use tumor samples from previous procedures. No new or additional procedures will be done for the purpose of this study.

The tumor samples will be sent to a lab for SmartMatch analysis. Once completed, the results will be shared with the patient and his/her local doctor. Together they can decide whether to incorporate the results into the treatment plan. It is important to know that the results may or may not be helpful.

There will only be one blood test for research. Blood and tissue samples collected may be used for additional analysis. Tumor tissue may be used to grow additional samples for further study. Participants will receive a pathology diagnosis and mutation profile generated by pathologists who specialize in CNS tumors.

The study team will seek updates on participant's health approximately every 6 months for 3 years. Tumor samples may also be collected from any additional surgery done at NIH during this time.

DETAILED DESCRIPTION:
Background:

* Primary central nervous system (CNS) tumors are uncommon and are mostly classified as rare diseases. Despite their low incidence, CNS cancers are associated with significant morbidity and mortality across all age groups.
* Treatment options for CNS tumors are limited, especially upon disease progression, largely due to the incomplete understanding of disease biology and the challenges in conducting clinical studies, given the rarity of these diseases.
* The traditional pathway for oncology drug development, involving several phases of clinical trials, can take many years to a decade and comes with a tremendously high financial cost. To overcome this challenge and speed up improving oncology patient care, drug repurposing has emerged as a useful approach.
* Real-time drug screening for rare brain tumors is advancing precision medicine by generating clinical trial concepts aimed at overcoming key challenges in brain tumor management. However, delayed turnaround times remain a significant limitation to their clinical utility.
* The Gujral lab at the Fred Hutchinson Cancer Center has developed SmartMatch, a cutting-edge artificial intelligence (AI)-driven system pharmacology-based platform to address the challenges in precision medicine. The platform allows the generation of drug response data using real-time tissue-based screening using freshly resected tumor or biopsy from a patient. The data collected is used to train a machine learning model, allowing precise prediction to a large panel of Food and Drug Administration (FDA)-approved drugs. This is a test that can be ordered by any physician in the US, and results are available upon request.

Objective:

-To determine the proportion of participants with advanced CNS tumors for whom SmartMatch drug screen analysis results are generated within 21 days from the time of tumor tissue acquisition

Eligibility:

* Participants >=15 years with advanced CNS tumors.
* Participants must have been scheduled for a brain tumor biopsy or resection planned to take place at NIH.

Design:

* Tumor and blood samples will be collected for multi-omic analysis.
* Fresh tumor samples will be used for drug screen analysis by SmartMatch.
* After initial sample collection, participants will be followed remotely every 6 (+/-3) months for 3 years.

ELIGIBILITY:
* INCLUSION CRITERIA
* Participants must have advanced CNS tumors confirmed by a documented pathology report, including:

  * recurrent isocitrate dehydrogenase (IDH)-wild-type high-grade glioma
  * recurrent IDH-mutant gliomas
  * other recurrent CNS tumors
* Participants must have been scheduled for a brain tumor biopsy or resection. Note: Scheduled brain tumor biopsy or resection must be at least 6 months after any previous radiation therapy, if applicable. All procedures are planned to take place at NIH.
* Age >= 15 years.
* Ability of participant, parent/guardian, or Legally Authorized Representative (LAR) to understand and sign a written informed consent document.

EXCLUSION CRITERIA

None.

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of participants with advanced CNS tumors for whom SmartMatch drug screen analysis results are generated within 21 days from the time of tumor tissue acquisition | 21 days from the time of tumor tissue acquisition
  Point estimates and 95% exact confidence intervals will be calculated using the Clopper-Pearson method

SECONDARY OUTCOMES:
To perform molecular profiling of advanced CNS tumors at disease progression. | End of Study
  Descriptive statistics will be used to summarize the molecular profiling results

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- [Background] Ostrom QT, Price M, Neff C, Cioffi G, Waite KA, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2015-2019. Neuro Oncol. 2022 Oct 5;24(Suppl 5):v1-v95. doi: 10.1093/neuonc/noac202. PMID 36196752
- [Background] Aldape K, Brindle KM, Chesler L, Chopra R, Gajjar A, Gilbert MR, Gottardo N, Gutmann DH, Hargrave D, Holland EC, Jones DTW, Joyce JA, Kearns P, Kieran MW, Mellinghoff IK, Merchant M, Pfister SM, Pollard SM, Ramaswamy V, Rich JN, Robinson GW, Rowitch DH, Sampson JH, Taylor MD, Workman P, Gilbertson RJ. Challenges to curing primary brain tumours. Nat Rev Clin Oncol. 2019 Aug;16(8):509-520. doi: 10.1038/s41571-019-0177-5. PMID 30733593
- [Background] Nishida-Aoki N, Bondesson AJ, Gujral TS. Measuring Real-time Drug Response in Organotypic Tumor Tissue Slices. J Vis Exp. 2020 May 2;(159). doi: 10.3791/61036. PMID 32420994
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002539-C.html